CLINICAL TRIAL: NCT00286507
Title: Full Thickness Macular Hole and Internal Limiting Membrane Peeling Study: Randomised Comparison of Macular Hole Surgery With or Without Internal Limiting Membrane Peeling
Brief Title: Full Thickness Macular Hole and Internal Limiting Membrane Peeling Study
Acronym: FILMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government); Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CZH/4/235
Record Dates: First submitted 2006-02-02; First posted 2006-02-03 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Stage 2 or 3 Full Thickness Macular Hole
Keywords: Full thickness macular hole; Internal limiting membrane (ILM); Vitreo retinal surgery; Vitrectomy
MeSH Terms: interventions — Vitrectomy; Gases

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- ILM peeling (Active Comparator): Combined cataract surgery (phacoemulsification and intraocular lens implantation) and pars plana vitrectomy with postoperative intraocular tamponade with gas, with ILM peeling
  Interventions: Procedure: Vitrectomy, post hyaloid detachment and gas injection with or without ILM peel.
- No ILM peeling (Active Comparator): combined cataract surgery (phacoemulsification and intraocular lens implantation) and pars plana vitrectomy with postoperative intraocular tamponade with gas without ILM peeling
  Interventions: Procedure: Vitrectomy, post hyaloid detachment and gas injection with or without ILM peel.

INTERVENTIONS:
Procedure: Vitrectomy, post hyaloid detachment and gas injection with or without ILM peel. — Combined cataract surgery (phacoemulsification and intraocular lens implantation) and pars plana vitrectomy with postoperative intraocular tamponade with gas, with or without ILM peeling

SUMMARY:
A macular hole is a fairly common problem in the retina and is an important cause of loss of central vision. The aim of this study is to determine whether, in patients with a stage 2 or 3 full thickness macular hole (FTMH), peeling a very fine, transparent tissue that covers the surface of the retina, called the internal limiting membrane (ILM) during surgery is superior to non-ILM peeling macular hole surgery. The main outcomes are improvement in vision, achievement of macular hole closure, need for re-operation, health related quality of life (HRQOL) and cost effectiveness.

DETAILED DESCRIPTION:
Idiopathic full-thickness macular hole (FTMH) is an important cause of loss of central vision, usually leading to severe visual impairment. Up to 20% of affected people will develop a FTMH in both eyes. There is uncertainty in the literature and among vitreo-retinal surgeons about the balance of potential benefits and adverse effects of ILM peeling in FTMH surgery for stage 2-3 holes.

FILMS is a randomised controlled trial (RCT) in patients with stage 2-3 FTMH less less than 18 months duration investigating whether ILM peeling improves the anatomical and visual outcome of macular hole surgery and the quality of life of patients with this retinal disease. Cost-effectiveness is also being addressed.

ELIGIBILITY:
Inclusion Criteria:

Idiopathic FTMH of stage 2-3, Duration of hole ≤18 months, Visual acuity equal to or worse than 20/40 in the study eye.

Exclusion Criteria:

Stage 1 or 4 FTMH, Stage 2-3 FTMH of > 18 months duration, Visual acuity >20/40 in study eye, FTMH related to high myopia (>6 dioptres), FTMH related to trauma, any other causes of decreased vision (ie corneal scarring, age-related macular degeneration, diabetic retinopathy, glaucoma if central and/or paracentral absolute visual field defects present), patient unable to understand English, patient unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2005-07; Primary Completion 2009-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study is the mean difference between treatment groups in the Early Treatment Diabetic Retinopathy Study (ETDRS) distance visual acuity score. | 6 months post surgery

SECONDARY OUTCOMES:
Secondary outcomes include anatomical closure, adverse events, re-operation, distance visual acuity (VA), near VA, contrast sensitivity, reading speed, costs to the health service and the participant and HRQOL. | 3, 6 and 24 months post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Noemi Lois, Principal Investigator — NHS Grampian
Locations (9):
- Ireland (2):
  - Royal Victoria Eye and Ear Hospital, Dublin
  - Waterford Regional Hospital, Waterford
- United Kingdom (7):
  - Aberdeen Royal Infirmary, Aberdeen
  - Bristol Eye Hospital, Bristol
  - Ninewells Hospital, Dundee
  - Gartnavel General Hospital, Glasgow
  - Royal Liverpool Hospital, Liverpool
  - Oxford Eye Hospital, Oxford
  - Sunderland Eye Infirmary, Sunderland

REFERENCES:
- [Derived] Lois N, Burr J, Norrie J, Vale L, Cook J, McDonald A, Boachie C, Ternent L, McPherson G; Full-thickness Macular Hole and Internal Limiting Membrane Peeling Study (FILMS) Group. Internal limiting membrane peeling versus no peeling for idiopathic full-thickness macular hole: a pragmatic randomized controlled trial. Invest Ophthalmol Vis Sci. 2011 Mar 1;52(3):1586-92. doi: 10.1167/iovs.10-6287. PMID 21051731
- [Derived] Lois N, Burr J, Norrie J, Vale L, Cook J, McDonald A; Full-Thickness Macular Hole and Internal Limiting Membrane Peeling Study (FILMS) Group. Clinical and cost-effectiveness of internal limiting membrane peeling for patients with idiopathic full thickness macular hole. Protocol for a randomised controlled trial: FILMS (Full-thickness Macular Hole and Internal Limiting Membrane Peeling Study). Trials. 2008 Nov 3;9:61. doi: 10.1186/1745-6215-9-61. PMID 18980675